CLINICAL TRIAL: NCT04578938
Title: Ketamine + Cognitive Training for Suicidality in the Medical Setting
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rebecca Price (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19100041 (Part 2); R01MH124983 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ketamine + Cognitive Training (Experimental)
  Interventions: Drug: Intravenous ketamine; Behavioral: Cognitive training
- Ketamine + Sham Training (Sham Comparator)
  Interventions: Drug: Intravenous ketamine; Behavioral: Sham Training
- No-infusion (TAU) + Cognitive Training (Active Comparator)
  Interventions: Behavioral: Cognitive training
- No-infusion (TAU) + Sham Training (Sham Comparator)
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Drug: Intravenous ketamine — Single subanesthetic infusion of ketamine (0.5mg/kg)
  Arms: Ketamine + Cognitive Training; Ketamine + Sham Training
Behavioral: Cognitive training — 8 sessions of computer-based cognitive training
  Arms: Ketamine + Cognitive Training; No-infusion (TAU) + Cognitive Training
Behavioral: Sham Training — 8 sessions of computer-based sham training
  Arms: Ketamine + Sham Training; No-infusion (TAU) + Sham Training

SUMMARY:
This project seeks to identify the acute and longer-term impact of a single dose of intravenous ketamine among suicidal patients referred for psychiatric consultation/liaison in the medical inpatient setting. The investigators will then test whether ketamine's rapid effects can be extended by introducing helpful information delivered by a computer-based training protocol. This work could ultimately lead to the ability to treat suicidality more efficiently and with broader dissemination by rapidly priming the brain for helpful forms of learning.

DETAILED DESCRIPTION:
NOTE: Edits were made to the outcome measures sections to improve clarity regarding the a priori analytic plan with respect to the "Time Frame" of measurements and to reduce redundancies. Timepoints that will be analyzed as trajectories over windows of time and measurements that will be analyzed as composites are now more clearly specified. The previous entries correctly identified all relevant measures and timepoints, but implied incorrectly that each timepoint/measure would be analyzed in isolation.

ELIGIBILITY:
Inclusion Criteria:

Participants who receive ketamine will:

1. be between the ages of 18 and 70 years
2. be a medical inpatient referred for psychiatric consultation/liaison due to suicidality and determined by psychiatric C/L to require follow-up psychiatric care (inpatient or outpatient)
3. possess a level of judgment and understanding sufficient to agree to all procedures required by the protocol and must sign an informed consent document
4. be deemed an appropriate and reasonable medical candidate for intravenous ketamine by a physician authorized to prescribe medication to the patient during inpatient hospitalization

Exclusion Criteria:

1. Presence of current/acute psychosis with significant thought disruption, mania, delirium, or dementia, or a diagnosis of developmental disorder with significant language and/or intellectual impairment
2. Mini-Mental State Exam (MMSE) < 21
3. Current pregnancy or breastfeeding
4. Reading level <5th grade as per WRAT-3 reading subtest AND patient declines to have all questionnaire items and task instructions read aloud to them at all assessment points
5. Past intolerance or hypersensitivity to ketamine or esketamine
6. Patients taking St John's Wort
7. Patients who have received ECT in the past 1 month prior to intake
8. Patients at ongoing risk for severe substance or alcohol withdrawal related issues (e.g., delirium tremens, severe opiate withdrawal) or who present with substance-induced psychosis
9. Arrested or incarcerated individuals brought in by the legal system for medical stabilization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicide Ideation | Trajectories from 24hrs through 1 month
  suicidal ideation/thoughts; range 0-38; high score=worse outcome
Montgomery Asberg Depression Rating Scale | Trajectories from 24hrs through 1 month
  depression severity; range 0-60; high score=worse outcome
Suicidal behaviors: medical chart review and Columbia Suicide Severity Rating Scale (CSSRS) | Trajectories from 24hrs through 12 months
  composite measure of # unique occurrences of any suicidal outcome (recorded via either measure) including: re-attempt, re-hospitalization for suicidality, suicide behaviors, or completed suicide

SECONDARY OUTCOMES:
Adult Suicide Ideation Questionnaire | Trajectories from 24hrs through 12 months
  suicidal ideation/thoughts; range 0-150; high score=worse outcome
Quick Inventory of Depressive Symptoms | Trajectories from 24hrs through 12 months
  Self-reported depression (range: 0-27; higher scores = worse outcome)
Scale for Suicide Ideation | Trajectories from 1 month through 12 months
  suicidal ideation/thoughts; range 0-38; high score=worse outcome
Montgomery Asberg Depression Rating Scale | Trajectories from 1 month through 12 months
  depression severity; range 0-60; high score=worse outcome

OTHER OUTCOMES:
Implicit Association Test | Trajectories from 24hrs through 1 week
  performance-based "target engagement" measure of suicidal cognition; range = -inf-inf; high score=worse outcome
Implicit Association Test | Trajectories from 1 week through 12 months
  performance-based "target engagement" measure of suicidal cognition; range = -inf-inf; high score=worse outcome
Acceptability: infusion | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Satisfaction: infusion | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Future likelihood of use: infusion | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Ease of use: Cognitive Training | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Helpfulness: Cognitive Training | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Satisfaction: Cognitive Training | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Future likelihood of use: Cognitive Training | Post-CT assessment (approximately +5 days post-randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
PROMIS Pain Intensity score | 24 hrs post-randomization
  PROMIS Pain Intensity Short Form scale T-score (range=0-100; higher score=worse pain)
PROMIS Pain Intensity score | Post-CT assessment (approximately +5 days post-randomization)
  PROMIS Pain Intensity Short Form scale T-score (range=0-100; higher score=worse pain)
PROMIS Neuropathic Pain Quality | 24 hrs post-randomization
  PROMIS Neuropathic Pain Quality scale T-score (range=0-100; higher score=worse pain)
PROMIS Neuropathic Pain Quality | Post-CT assessment (approximately +5 days post-randomization)
  PROMIS Neuropathic Pain Quality scale T-score (range=0-100; higher score=worse pain)
PROMIS Nociceptive Pain Quality | 24 hrs post-randomization
  PROMIS Nociceptive Pain Quality scale T-score (range=0-100; higher score=worse pain)
PROMIS Nociceptive Pain Quality | Post-CT assessment (approximately +5 days post-randomization)
  PROMIS Nociceptive Pain Quality scale T-score (range=0-100; higher score=worse pain)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca B Price, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No